CLINICAL TRIAL: NCT05969977
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Combined Single and Multiple Ascending Dose Study of PPI-1011 in Subjects to Assess Safety, Tolerability, and Pharmacokinetics
Brief Title: A First-in-Human Phase 1 Study of Plasmalogen Precursor PPI-1011 in Healthy Adult Volunteers to Assess Safety, Tolerability, and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MED-LIFE DISCOVERIES LP (Industry)
Collaborators: BioPharma Services Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLD-CT-1.1
Record Dates: First submitted 2023-06-11; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Rhizomelic Chondrodysplasia Punctata
Keywords: Phase 1; Healthy Adult Volunteer; RCDP; Plasmalogen; Rhizomelic Chondrodysplasia Punctata
MeSH Terms: conditions — Chondrodysplasia Punctata, Rhizomelic | interventions — PPI-1011

STUDY DESIGN:
Intervention Model Description: The study consists of 5 planned single-dose cohorts (n = 8 per cohort, total randomized 6 active: 2 placebo) with sentinel design followed by 2 multiple-dose cohorts (n = 8 per cohort, total randomized 6 active: 2 placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPI-1011 (Experimental): Single Ascending: PPI-1011 at 10, 25, 50, 75 and 100 mg/kg. Multiple Dose: PPI-1011 dose to be based on SAD; duration 14 days; one dose daily.
  Interventions: Drug: PPI-1011
- Placebo (Placebo Comparator): Placebo arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPI-1011 — PPI-1011 is a liquid oil with light yellow to amber color, clear to slightly opalescent and flows readily at room temperature. It is insoluble in water and miscible with dichloromethane and liquid coconut oil. It is a synthetic glycerolipid derivative, comprised of an assembly of naturally-occurring products including glycerol backbone, an ether-linked hexadecyl group at sn1 position, an all-cis-4, 7, 10, 13, 16, 19-docosahexaenoyl group at sn2 position, and a lipoyl group at sn3 position. It was designed as a plasmalogen precursor and is similar in structure to naturally occurring alkyl-diacyl lipids with the primary difference being the presence of a lipoic acid moiety at the sn3 position. PPI-1011 is formulated in liquid coconut oil containing 0.1% 1-thioglycerol as an antioxidant.
  Arms: PPI-1011
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
PPI-1011 is being developed as a docosahexaenoic acid (DHA) containing plasmalogen precursor with good long-term stability, specifically for the treatment of rhizomelic chondrodysplasia punctata (RCDP), which is an ultra rare type of peroxisomal biogenesis disorder (PBD). The goal of treatment with PPI-1011 is to increase the levels of plasmalogens within circulation and tissues, with the hope that this will normalize plasmalogen levels in the body and result in clinical improvement to patients. The present study is a first-in-human (FIH), phase 1, randomized, double-blind, placebo-controlled, dose-escalation study to assess the safety, tolerability and pharmacokinetics (PK) of single and multiple ascending doses of PPI-1011 administered orally to healthy subjects. The study consists of 5 planned single-dose cohorts (n = 8 per cohort, total randomized 6 active: 2 placebo) with sentinel design. Following a review of the safety and PK data by the safety review committee and submission to Health Canada the study will be expanded to include 2 planned multiple-dose cohorts (n = 8 per cohort, total randomized 6 active: 2 placebo).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, first-in-human (FIH) study of PPI-1011 in healthy male and non-pregnant, non-lactating female volunteers. The study will consist of two parts: single ascending dose (SAD) and multiple ascending dose (MAD). The study will evaluate the safety, tolerability and PK in 5 planned SAD cohorts with sentinel design (n=8 per cohort, total randomized 6 active: 2 placebo) and 2 planned MAD cohorts (n=8 per cohort, total randomized 6 active: 2 placebo). Based on accumulating data, additional single-dose and/or a multiple-dose cohort(s) (n=8 per cohort) may be added to better assess the safety, tolerability, or PK profile of PPI-1011 to meet study objectives and try to determine the maximum tolerated dose.

A sentinel dose in 2 participants (1:1 PPI-1011: placebo) will be performed in each single-dose cohort to evaluate the safety and tolerability at planned doses. Additional cohort(s) will be dosed in case a different dose(s) is required based upon the emerging safety and PK data from the main cohort(s) to provide better assessment for the safety, tolerability, or PK of PPI-1011. A sentinel design may not be applicable when a cohort with the same or a higher drug exposure has already been evaluated.

Single Ascending Dose (SAD):

The 5 planned single-dose levels are:

Cohort A 10 mg/kg PPI-1011 or Placebo Cohort B 25 mg/kg PPI-1011 or Placebo Cohort C 50 mg/kg PPI-1011 or Placebo Cohort D 75 mg/kg PPI-1011 or Placebo Cohort E 100 mg/kg PPI-1011 or Placebo

Dose levels may be changed and/or additional cohorts may be added based on emerging safety and PK data. Subjects enrolled in the single-dose treatment cohorts will receive a single dose of the study drug (PPI-1011 or placebo) orally on Day 1.

A period of at least 24 hours will be required between administering study drug to the first 2 subjects (1 active, 1 placebo) and the 6 remaining subjects (5 active, 1 placebo) in the cohort. If no major safety concerns are observed following 24 hours of observation, dosing of the remaining 6 participants in that cohort may proceed. The dose-escalation may proceed after the Safety Review Committee review of the blinded safety data up to at least Day 3 from all participants in the preceding single-dose cohort. The dose escalation decision will be based on safety evaluation for an acceptable safety profile as determined by the SRC.

Cohorts A, B, C, D, and E will be dosed in a non-fasting state.

Multiple Ascending Dose (MAD):

The 2 planned multiple-dose levels are:

Cohort AA:

Study Drug Dose*: TBD mg/kg PPI-1011 or Placebo Dosing Regimen*: 1 x TBD mg/kg every 24 hours Duration (Days): 14 Total Dose (mg/kg): TBD

Cohort BB:

Study Drug Dose*: TBD mg/kg PPI-1011 or Placebo Dosing Regimen*: 1 x TBD mg/kg every 24 hours Duration (Days): 14 Total Dose (mg/kg): TBD

Cohorts AA and BB will be dosed in a non-fasting state.

*MAD dosing levels will be decided after review of the safety and PK data from the SAD cohorts. The SRC will propose doses, which will be submitted to Health Canada, together with the safety and PK data from the SAD. Dose levels may be further adjusted based on emerging safety and PK data from MAD cohorts.

Subjects enrolled in the multiple-dose treatment cohorts will receive oral doses of the study drug (PPI-1011 or placebo) once daily at 24-hour intervals. Thus, the total number of doses subjects will receive in a MAD cohort will be up to 14 doses. The doses for these cohorts will be selected after review of the blinded safety and PK data by the SRC and submitted to Health Canada. The dose in the MAD will not exceed the doses tested in the SAD.

Treatment Phases:

Single-Dose Cohorts (In-Clinic):

Participants will check in on Day -1. On Day 1, participants will receive a single dose of PPI-1011 or placebo. Participants will remain confined in the clinic from Day -1 until Day 2 (at least 36 hours after dosing). Participant can stay longer in the clinic if deemed necessary upon the Investigator's discretion.

Single-Dose Cohorts (Outpatient Visits):

After completing the in-house confinement period, participants will return to the clinic for an outpatient visit on Day 3, Day 4, Day 5 and Day 6.

Multiple-Dose Cohorts (In-Clinic):

Participants will check in on Day -1. Participants will receive oral doses of PPI-1011 or placebo from Day 1 to Day 14. Participants will remain confined in the clinic from Day -1 through Day 15 (at least 36 hours after the last dose). Participant can stay longer in the clinic if deemed necessary upon the Investigator's discretion.

Multiple-Dose Cohorts (Outpatient Visits):

After completing the confinement period, participants will return to the clinic for an outpatient visit on Day 16, Day 17, Day 18 and Day 19.

Study Numbers:

Fifty-six (56) healthy volunteers are planned to be enrolled in this study. Forty (40) subjects will be enrolled in the SAD portion of the study and 16 subjects will be enrolled in the MAD portion (n=8 per cohort). For SAD cohorts, each cohort will enroll a minimum of 3 subjects of each sex, with at least 2 males and 2 females randomized to the active treatment. The same may be implemented for MAD cohorts based on emerging safety and PK data.

Additional subjects (in single [n=8] or multiple dose [n=8] cohorts) may be added to better assess the safety, tolerability, or PK of PPI-1011 to meet study objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking (for at least 6 months prior to first study drug administration) male, and non-pregnant and non-lactating female (including post-menopausal and surgically sterile female) volunteers, 18-65 years of age, inclusive at the time of informed consent.

   * Post-menopausal for at least 1 year [confirmed by FSH (16-157 IU/L) and 17β-estradiol (<202 pmol/L) levels]

     * Surgically sterile (Partial or total hysterectomy, bilateral oophorectomy, bilateral salpingo-oophorectomy) for at least 6 months [confirmed by medical/operative report or if medical/operative report is not available by FSH and 17β-estradiol tests, if applicable].
2. Body mass index (BMI) that is within 18.5 - 30.0 kg/m2, inclusive, and subject weighs no more than 91.0 kg.
3. Healthy, according to the medical history, ECG, vital signs, laboratory results and physical examination as determined by the PI/Sub-Investigator.
4. Systolic blood pressure between 95-140 mmHg, inclusive, and diastolic blood pressure between 55-90 mmHg, inclusive, oxygen saturation level between 95% and 100%, inclusive, and heart rate between 55-100 bpm, inclusive, unless deemed otherwise by the PI/Sub-Investigator.
5. Clinical laboratory values within BPSI's most recent acceptable laboratory test range, and/or values are deemed by the PI/Sub-Investigator as "Not Clinically Significant".
6. Ability to comprehend and be informed of the nature of the study, as assessed by BPSI staff. Capable of giving written informed consent prior to any study related procedure. Must be able to communicate effectively with clinic staff.
7. Ability to fast for at least 10 hours and consume standard meals.
8. Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements.
9. Agree not to have a tattoo or body piercing until the end of the study.
10. Agree not to receive COVD-19 vaccination from 7 days prior to first study drug administration until 7 days after the last study drug administration or the last procedure in the study, whichever is later.
11. Agree not to receive a vaccination (live attenuated vaccine) during the study and until 60 days after the study has ended (last study procedure)
12. Female subjects must be non-pregnant and non-lactating and fulfil at least one of the following:

    * Be surgically sterile for a minimum of 6 months (achieved through partial or total hysterectomy, bilateral oophorectomy, or bilateral salpingectomy; note that tubal ligation is not considered a method of permanent sterilization).
    * Post-menopausal for a minimum of 1 year [confirmed by FSH (16-157 IU/L) and 17β-estradiol (<202 pmol/L) levels]) (post-menopausal is defined as 12 consecutive months with no menses without an alternative medical cause).
    * Agree to avoid pregnancy and use an acceptable highly effective method of contraception with male sexual partners from at least 30 days prior to the study until at least 30 days after the study has ended (last study procedure).

    Medically acceptable methods of contraception include oral contraceptives, hormonal patch, implant or injection, hormonal or non-hormonal intrauterine device (IUD) combined with a barrier method (male or female condom, diaphragm with spermicide, or cervical cap with spermicide) or double barrier methods (male condom in conjunction with diaphragm and spermicide, male condom in conjunction with cervical cap and spermicide). Complete abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the subject.

    If a subject becomes pregnant during her participation in the study and for 30 days after she has completed her last study study procedure, she must inform BPSI staff immediately.
13. Males who are not vasectomized for at least 6 months prior to dosing and are able to father children must agree to use an acceptable highly effective method of contraception with female sexual partners of childbearing potential and not donate sperm during the study and for at least 30 days after the last study drug administration.

Medically acceptable methods of contraception include using a condom with a female sexual partner of childbearing potential who is using oral contraceptives, hormonal patch, implant or injection, IUD or system, or diaphragm with spermicide. Complete abstinence as a method of contraception is acceptable if it is in line with the preferred and usual lifestyle of the subject.

If a subject's partner becomes pregnant during his participation in the study and for 30 days after he has completed his last study drug administration, he must inform BPSI staff immediately.

Exclusion Criteria:

1. Known history or presence of any clinically significant hepatic, renal/genitourinary, gastrointestinal, cardiovascular, cerebrovascular, pulmonary, endocrine, immunological, musculoskeletal, neurological, psychiatric, dermatological or hematological disease or condition unless determined as not clinically significant by the PI/Sub-Investigator.
2. Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g., chronic diarrhea, inflammatory bowel disease), unresolved gastrointestinal symptoms (e.g., diarrhea, vomiting), or other conditions known to interfere with the absorption, distribution, metabolism or excretion of the drug experienced within 7 days prior to first study drug administration, as determined by the PI/Sub-Investigator.
3. Presence of any clinically significant illness within 30 days prior to first dosing, as determined by the PI/Sub-Investigator.
4. Presence of any significant physical or organ abnormality as determined by the PI/Sub-Investigator.
5. A known history or positive test result for human immunodeficiency virus (HIV), chronic Hepatitis B surface antigen, or Hepatitis C.
6. A positive test result for drugs of abuse/recreational drugs (marijuana, amphetamines, barbiturates, cocaine, opiates, phencyclidine and benzodiazepines), alcohol test and cotinine. Positive pregnancy test for female subjects of childbearing potential.
7. Known history or presence of:

   * Alcohol abuse or dependence within one year prior to first study drug administration;
   * Drug abuse or dependence;
   * Known hypersensitivity or idiosyncratic reaction to PPI-1011, its excipients (e.g., liquid coconut oil, 1-thioglycerol etc), and/or related substances;
   * Food allergies;
   * Presence of any dietary restrictions unless deemed by the PI/Sub-Investigator as "Not Clinically Significant";
   * Severe allergic reactions (e.g. anaphylactic reactions, angioedema).
   * Intolerance to and/or difficulty with blood sampling through venipuncture.
   * Abnormal diet patterns (for any reason) during the four weeks preceding the study, including fasting, high protein diets etc.

10. Individuals who have donated, in the days prior to first study drug administration:

* 50-499 mL of blood in the previous 30 days;
* 500 mL or more in the previous 56 days. 11. Donation of plasma by plasmapheresis within 7 days prior to first study drug administration.

  12. Individuals who have participated in another clinical trial or who received an investigational drug within 30 days prior to first study drug administration.

  13. Use of any lipid lowering drug/agent including hydroxymethylglutaryl (HMG) CoA reductase inhibitors (Statins), cholesterol absorbing inhibitors (Ezetimibe), fibric acid derivatives (Fibrates), bile acid sequestrants, PCSK9 inhibitors, and nicotinic acid within 30 days prior to first study drug administration and for the duration of the study.

  14. Use of of any supplements containing DHA, fish oil, krill oil, plasmalogen extract or scallop extracts within 30 days prior to first study drug administration and for the duration of the study.

  15. Use of any supplements containing lipoic acid within 30 days prior to first study drug administration and for the duration of the study.

  16. Use of any prescription medication within 14 days prior to first study drug administration (except for accepted methods of contraception).

  17. Use of any over-the-counter medications (including oral multivitamins, herbal and/or dietary supplements) within 14 days prior to first study drug administration (except for accepted methods of contraception).

  18. Consumption of food or beverages containing grapefruit and/or pomelo within 10 days prior to first study drug administration.

  19. Consumption of food or beverages containing caffeine/methylxanthines, poppy seeds and/or alcohol within 48 hours before dosing.

  20. Individuals having undergone any major surgery within 6 months prior to the start of the study, unless deemed otherwise by PI/Sub-Investigator.

  21. Have any other conditions that, in the opinion of the Investigator or Sponsor, would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the study.

  22. Difficulty with swallowing the study drug (oral solution). 23. Have tongue piercings and/or mouth jewelry. 24. Women who are pregnant or lactating. 25. Unable or unwilling to provide informed consent 26. Have had a tattoo or body piercing within 30 days prior to first study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events as assessed by the CTCAE scale | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the last dose in multiple ascending dose subjects.
  Emergence of adverse events will be documented for incidence, severity and duration and rated according to the CTCAE criteria.

SECONDARY OUTCOMES:
Pharmacokinetics-AUC | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the last dose in multiple ascending dose subjects.
  Characterize the pharmacokinetics of PPI-1011 using the AUC
Pharmacokinetics-Cmax | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the last dose in multiple ascending dose subjects.
  Characterize the pharmacokinetics of PPI-1011 using the peak serum concentration (Cmax)
Pharmacokinetics-Tmax | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the last dose in multiple ascending dose subjects.
  Characterize the pharmacokinetics of PPI-1011 by determining the time of the maximum serum concentration (Tmax).
Pharmacokinetics-T1/2 | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the last dose in multiple ascending dose subjects.
  Characterize the pharmacokinetics of PPI-1011 by determining the terminal half-life in serum (T1/2).
Pharmacokinetics-λ | Up to 6 days post-dose in single ascending dose subjects and up to 7 days post the lst dose in multiple ascending dose subjects.
  Characterize the pharmacokinetics of PPI-1011 by determining the terminal elimination rate constant (λ) in serum.
Pharmacokinetics-CL/F | Up to 6 days post-dose in single ascending dose subjects
  Characterize the pharmacokinetics of PPI-1011 by determining the apparent total body clearance calculated after a single extravascular administration (CL/F).
Pharmacokinetics-Vd/F | Up to 6 days post-dose in single ascending dose subjects
  Characterize the pharmacokinetics of PPI-1011 by determining the apparent volume of distribution after oral administration based on the terminal phase calculated after a single extravascular administration (Vd/F).
Pharmacokinetics-Accumulation ratio (AR) | Up to 24 hrs after the final dose in multiple ascending dose participants.
  Characterize the pharmacokinetics of PPI-1011 by determining the accumulation ratio of PPI-1011 following 14 days of oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Smith, PhD, Study Director — MED-LIFE DISCOVERIES LP
Locations (1):
- Biopharma Services Inc., Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No